CLINICAL TRIAL: NCT01683084
Title: Study of the Effectiveness of Telmisartan in Slowing the Progression of Abdominal Aortic Aneurysms
Acronym: TEDY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: Medtronic (Industry); James Cook University, Queensland, Australia (Other)
Responsible Party: Principal Investigator, Ronald L. Dalman, MD, Chidester Professor of Surgery and Chief, Stanford Vascular Surgery, Palo Alto Veterans Institute for Research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAL0041ARG; 22647 (Other: Stanford IRB)
Record Dates: First submitted 2012-09-05; First posted 2012-09-11 (Estimated); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Abdominal Aortic Aneurysm; AAA; telmisartan
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Telmisartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Telmisartan (Active Comparator): One 40mg telmisartan pill given once daily for 24 months
  Interventions: Drug: Telmisartan
- Placebo (Placebo Comparator): One 40mg placebo pill given once daily for 24 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Telmisartan
  Arms: Telmisartan
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if telmisartan is effective in slowing the progression of abdominal aortic aneurysms and reducing circulating concentrations of Abdominal Aortic Aneurysms (AAA) biomarkers.

DETAILED DESCRIPTION:
Currently, the only management options for AAA are surgical (open or endovascular) based on ongoing follow-up with imaging at regular intervals. Telmisartan is currently approved for use in the United States by the Food and Drug Administration for management of hypertension. If telmisartan is found to be effective in slowing the progression of abdominal aortic aneurysms, this would provide a new treatment option for patients with AAA disease.

ELIGIBILITY:
Inclusion Criteria:

* 50-85 years of age and able to provide written informed consent
* AAA measuring a maximum diameter of 3.5-4.9 cm on CTA or ultrasound
* Stable medication regime for the last six months
* No current indication for AAA repair according to the treating physician or expectation that this will be revised within the next year
* High likelihood of compliance with treatment over 24 months

Exclusion Criteria:

* Renal impairment (i.e. creatinine >1.5x upper limit of normal [ULN])
* Known significant renal stenosis (>70%) of one or both renal arteries
* Chronic liver disease (i.e. cirrhosis or hepatitis) or abnormal liver function (i.e. ALT 1.5xULN)
* Electrolyte imbalance
* Active gout
* Current or planned usage of an AT1 blocker or ACE inhibitor
* Previous abdominal aortic surgery
* Currently pregnant or intend to become pregnant

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-09-19 (Actual); Primary Completion 2018-11-10 (Actual); Study Completion 2018-11-10 (Actual)

PRIMARY OUTCOMES:
Rate of AAA growth assessed by total infrarenal aortic volume measured on computed tomography angiography (CTA) | Patients will be followed for two years following enrollment, with AAA growth determined by comparing total AAA volume at baseline and at two years between control and treatment groups.

SECONDARY OUTCOMES:
Change in maximum infrarenal AAA diameter and aortic distensibility on repeat ultrasound | Comparison between two groups at baseline and two years.
  Interval assessments of ultrasound-determined diameter will also be performed to reduce the variability of individual ultrasound-derived aortic diameter measurements.
Change in circulating concentrations of AAA biomarkers (serum OPG, OPN, MMP-9 and TGFB-1) on repeated samples | Comparison between baseline and 2 years (24 months) following enrollment
Quality of life assessed by the 12-item Assessment of Quality of Life (AQoL) | Comparison between baseline and 24 months between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald L Dalman, M.D., Principal Investigator — PAIRE: Stanford University, VA Palo Alto Health Care System
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

REFERENCES:
- [Background] Golledge J, Tsao PS, Dalman RL, Norman PE. Circulating markers of abdominal aortic aneurysm presence and progression. Circulation. 2008 Dec 2;118(23):2382-92. doi: 10.1161/CIRCULATIONAHA.108.802074. No abstract available. PMID 19047592
- [Derived] Golledge J, Pinchbeck J, Tomee SM, Rowbotham SE, Singh TP, Moxon JV, Jenkins JS, Lindeman JH, Dalman RL, McDonnell L, Fitridge R, Morris DR; TEDY Investigators. Efficacy of Telmisartan to Slow Growth of Small Abdominal Aortic Aneurysms: A Randomized Clinical Trial. JAMA Cardiol. 2020 Dec 1;5(12):1374-1381. doi: 10.1001/jamacardio.2020.3524. PMID 32845283
- [Derived] Xuan H, Xu B, Wang W, Tanaka H, Fujimura N, Miyata M, Michie SA, Dalman RL. Inhibition or deletion of angiotensin II type 1 receptor suppresses elastase-induced experimental abdominal aortic aneurysms. J Vasc Surg. 2018 Feb;67(2):573-584.e2. doi: 10.1016/j.jvs.2016.12.110. Epub 2017 Apr 20. PMID 28434702
- [Derived] Morris DR, Cunningham MA, Ahimastos AA, Kingwell BA, Pappas E, Bourke M, Reid CM, Stijnen T, Dalman RL, Aalami OO, Lindeman JH, Norman PE, Walker PJ, Fitridge R, Bourke B, Dear AE, Pinchbeck J, Jaeggi R, Golledge J. TElmisartan in the management of abDominal aortic aneurYsm (TEDY): The study protocol for a randomized controlled trial. Trials. 2015 Jun 17;16:274. doi: 10.1186/s13063-015-0793-z. PMID 26081587